CLINICAL TRIAL: NCT00252395
Title: Effects of Electronic Prescribing on Safety and Quality in Hospital-Based Ambulatory Are: a Randomised Controlled Trial
Brief Title: Evaluation of Electronic Prescribing in Hospital Ambulatory Care Clinics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Health Canada (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: S&W e-RX; 6804-15-2003/5590024
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2005-11-11 (Estimated); Status verified 2005-11

CONDITIONS: Electronic Prescribing
Keywords: medication error; electronic prescribing; patient safety

INTERVENTIONS:
Device: PDA-based Electronic Prescribing Software

SUMMARY:
All reliably evaluated POE systems to date have been desktop computer based, but now there is widespread use and acceptance among physicians of PDA devices for a variety of purposes. Clinicians report that drug information on a PDA improved their access to information and efficiency while reducing their self perceived error rates6. The use of these devices for information retrieval in clinical settings is expected to grow as wireless communication becomes more ubiquitous and as more applications become available6,7. During the past decade there has been a growing awareness of several issues aimed at promoting safer health care for our patients - point of care information technology is one of the keys.

To this end we have worked with a Canadian company, Drugmagnet, to develop and implement PDA-based electronic prescribing system within a major Canadian academic health centre. This is a cluster randomised trial, in which access to and use of the e-prescribing system is switched on and off for randomly chosen weeks, thus time serves as the randomized element.

ELIGIBILITY:
Inclusion Criteria:

* active staff physician at Sunnybrook & Women's College HSC

Exclusion Criteria:

* inadequate prescribing practice (minimum number)

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-08; Study Completion 2006-08

PRIMARY OUTCOMES:
Total prescribing error, as measured by the number of call backs received from pharmacists.

SECONDARY OUTCOMES:
a) Interactions
b) Dosing and route of administration errors
c) Pack errors
d) Legibility errors

CONTACTS AND LOCATIONS:
Overall Officials: Merrick F Zwarenstein, MBBCH, Study Director — Institute for Clinical Evaluative Science; William J Sibbald, MD, MPH, Principal Investigator — Sunnybrook & Women's College Health Sciences Centre
Locations (1):
- Sunnybrook & Women's College Health Science Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dainty KN, Adhikari NK, Kiss A, Quan S, Zwarenstein M. Electronic prescribing in an ambulatory care setting: a cluster randomized trial. J Eval Clin Pract. 2012 Aug;18(4):761-7. doi: 10.1111/j.1365-2753.2011.01657.x. Epub 2011 Mar 18. PMID 21414109
- [Derived] Zwarenstein MF, Dainty KN, Quan S, Kiss A, Adhikari NK. A cluster randomized trial evaluating electronic prescribing in an ambulatory care setting. Trials. 2007 Oct 3;8:28. doi: 10.1186/1745-6215-8-28. PMID 17915028